CLINICAL TRIAL: NCT04667715
Title: A Pivotal Study to Evaluate the Safety and Effectiveness of Exablate Model 4000 Using Microbubble Resonators to Temporarily Mediate Blood-Brain Barrier Disruption (BBBD) in Subjects With Suspected Infiltrating Glioma
Brief Title: Safety and Effectiveness of Blood-Brain Barrier Disruption (BBBD) in Subjects With Suspected Infiltrating Glioma
Acronym: BBBD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company decision to switch to other trials
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT011
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Independent Reviewers (neurosurgeon/neuroradiologist), functioning as an Imaging Review Core Lab, will be blinded to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Exablate Test Arm (Active Comparator): Subjects will undergo ExAblate BBBD prior to their standard of care tumor removal
  Interventions: Device: Exablate BBBD
- Control Test Arm (No Intervention): Subjects will undergo their standard of care tumor removal

INTERVENTIONS:
Device: Exablate BBBD — Blood brain barrier disruption using ExAblate Type 2 device using microbubble resonators
  Arms: Exablate Test Arm

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of using the Exablate Type 2 system using microbubble resonators (Exablate Test Arm) to disrupt the Blood-Brain Barrier for the purpose of temporarily transforming, and thereby 'marking', regions of infiltrating gliomas prior to planned surgical resection, for the purpose of improving tumor visualization during the surgery to achieve a greater proportion of subjects who receive a Gross Total Resection (GTR) per plan compared to those not undergoing a BBBD procedure prior to resection (Control Arm).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening to determine eligibility for study entry. Patients who meet the eligibility requirements will be randomized in a 2:1 ratio to Exablate Test Arm and to Control Arm, respectively. The following assessments will occur:

1. Pre-surgical planning and Post-surgical visit MRI exams with and without contrast will be collected for evaluation by the study core lab; Any return to surgery for additional resection will be captured
2. All subjects will be seen at ~Week 2, and ~4-Weeks post resection for physical and neurological exams and to assess for complications or adverse events. These visits should coincide with standard (Neuro-oncology) care following resection.
3. Long-term outcomes will be collected during standard of care Neuro-oncology care follow-up visits for up to 2 years post resection; standard of care MRIs and RANO assessments will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female between 21-85 years of age who are able and willing to give informed consent
2. Subjects with suspected Grade II, III or IV infiltrating glioma (IG) on pre-operative brain imaging scans who have a non-enhancing component and are planned for surgical resection.
3. Karnofsky Performance Score 70-100
4. Able to communicate sensations during the Exablate BBBD procedure

Exclusion Criteria:

1. Tumor originating from the deep midline, thalamus, midbrain, cerebellum or brainstem.
2. Multifocal tumors
3. MRI or clinical findings of:

   1. Active or chronic infection(s) or inflammatory processes
   2. Acute or chronic hemorrhages, specifically any lobar microbleeds, and no siderosis, amyloid angiopathy, or macro-hemorrhages
   3. Intracranial thrombosis, vascular malformation, cerebral aneurysm or vasculitis
4. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
5. MR non-compatible metallic implants in the skull or the brain or the presence of unknown MR unsafe devices
6. Significant cardiac disease or unstable hemodynamic status

   1. Documented myocardial infarction within six months of enrollment
   2. Unstable angina on medication
   3. Unstable or worsening congestive heart failure
   4. Left ventricular ejection fraction below the lower limit of normal
   5. History of a hemodynamically unstable cardiac arrhythmia
   6. Cardiac pacemaker
   7. Patient has right-to-left, bidirectional, or transient right-to-left cardiac shunts
   8. Subjects with relative contraindications to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation,
   9. Perflutren sensitivity or allergy ii. QT prolongation observed on screening ECG (QTc > 450 for men and >470 for women)
7. Uncontrolled hypertension (systolic > 180 and diastolic BP > 120 on medication)
8. Unable to discontinue use of anti-coagulant/antiplatelet therapy as per local standard.
9. History of a liver disease, bleeding disorder, coagulopathy or a history of spontaneous hemorrhage or evidence of increased risk of bleeding
10. Abnormal coagulation profile (Platelets < 80,000), PT (>14) or PTT (>36), and INR > 1.3.
11. Large lacunar lesions that cannot be navigated around
12. Known cerebral or systemic vasculopathy
13. Significant depression and at potential risk of suicide
14. Known sensitivity/allergy to gadolinium, or other intravascular contrast agents
15. Active seizures despite medication treatment (defined as >1 seizure per week) which could be worsened by disruption of the blood brain barrier
16. History of anaphylactic shock
17. Active drug or alcohol disorder which have a higher risk for seizures, infection and/or poor executive functioning
18. Positive HIV status, which can lead to increased entry of HIV into the brain parenchyma leading to HIV encephalitis
19. Potential blood-borne infections which can lead to increased entry to brain parenchyma leading to meningitis or brain abscess
20. Any contraindications to MRI scanning,
21. Impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
22. Severe Respiratory Illness
23. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device
24. Pregnancy or Lactation

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-23 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Overall safety of the Exablate BBBD procedure itself as measured through the collection of adverse events | Approximately 2 months
  Safety of the Exablate BBBD procedure will be evaluated by patient examination and post-procedure MRI exams assessing changes in the treated region. Adverse events will be reported by the Investigator and monitored in both treatment arms.
Effectiveness of BBBD as determined by the proportion of subjects in whom a GTR is acheived | MRI 72 hours post resection
  The proportion of subjects in whom a gross total resection (actual versus planned) is achieved as measured on post-operative imaging compared to pre-resection imaging

SECONDARY OUTCOMES:
Confirmation of accuracy of Exablate BBBD targeting | MRI immediately after the ExAblate procedure
  Confirmation that new BBBD by contrast enhancement in a previously non-enhancing area overlies the intended target for BBBD. (ExAblate arm only)
Return Rate for Second Surgery for Completion of Resection | Approximately 2 months
  Comparison of the Return Rate between the two treatment arms.

OTHER OUTCOMES:
Evaluation of circulating tumor biomarkers | pre- and post-BBBD procedure
  Collection of blood for evaluation of circulating tumor biomarkers (e.g. circulating tumor DNA [ctDNA])

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Woodworth, MD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No